CLINICAL TRIAL: NCT04384029
Title: Retrospective Observational Study to Compare the Short, Mid- and Long-term Prognosis and Outcomes of SRAS-CoV-2 Infected Hospitalized Patients With Cardiovascular Disease (CVD) to SARS-CoV-2 Infected Hospitalized Patients Without CVD: The Geneva Covid-19 CVD Study
Brief Title: The Geneva Covid-19 CVD Study
Status: Completed | Type: Observational
Sponsor: François MACH (Other)
Responsible Party: Sponsor-Investigator, François MACH, Professor François MACH, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: CCER-2020-00610
Record Dates: First submitted 2020-04-20; First posted 2020-05-12 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: COVID; CVD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Covid-19 + patients — all the patients hospitalized in Geneva and SARS-Cov2 positive

SUMMARY:
In this study, the investigators propose to analyse the clinical data of all patients admitted in Geneva University Hospitals (HUG) or in a care center in Geneva who are diagnosed with COVID-19. CVD being one of the most important risk factors for developing a severe form of the disease, the investigators will explore the prognosis and clinical outcomes of those patients according to their CVD history as well as newly onset CVD during hospitalization. Moreover, as further evidence is needed on the use of renin-angiotensin-aldosterone system (RAAS) inhibitors for SARS-CoV-2 infected patients, the investigators will study prognosis and outcomes according to the patients' medications. Finally, the investigators propose to evaluate hospital length of stay and cost. The aim, therefore, is to collect information and scientific evidence from patients hospitalized and diagnosed positive for COVID-19, in order to evaluate if previous (or newly onset) CVD may influence outcomes and costs.

DETAILED DESCRIPTION:
Hypothesis:

COVID-19+ hospitalized patients with preexisting CVD or newly onset CVD at time of hospitalization have different clinical outcomes compared to those without CVD and COVID-19+.

Objectives:

The primary aim of this study is to gather observational data, starting from February 1st 2020 until the end of the pandemic, to compare clinical outcomes COVID+ hospitalized patients at HUG or in a care center in Geneva with pre-existing or newly onset CVD, to COVID+ hospitalized patients at HUG or in a care center in Geneva without pre-existing CVD.

The secondary aims of this study are:

* To determine the association between COVID-19 disease and CVD, based on: age, previous CV diseases, CV risks factors, CV medications (e.g. ACE Inhibitors or angiotensin II receptor antagonists)
* To explore CVD profiles that may influence COVID-19 disease outcomes
* To determine the cause of death in CVD patients (either with preexisting CVD or newly diagnosed with CVD)
* To understand the vulnerability of the myocardium (new event of either heart failure, acute coronary syndrome, arrhythmia, myocarditis) in patients with COVID-19 disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥18 years of age.
* Patient diagnosed SARS-CoV-2 positive at time of hospitalization.
* In case of the subject accepting the follow-up at 30 days and 1 year, Signed Patient Informed Consent (PIC) form

Exclusion Criteria:

* Patients unwilling to provide informed consent for the follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational study will include male and female patients hospitalized with a COVID+ diagnosis at the HUG or in a care center in Geneva.
Sampling Method: Non-Probability Sample
Enrollment: 1927 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
mobidity discharge | 0 days after hospitalization
  To compare morbidity during hospital stay in COVID-19+ patients with or without preexisting CVD.
mobidity at 30 days | 30 days after hospitalization
  To compare morbidity 30 days after hospitalization in COVID-19+ patients with or without preexisting CVD.
mobidity 1 year after hospitalization | 1 year after hospitalization
  To compare morbidity 1 year after hospitalization stay in COVID-19+ patients with or without preexisting CVD.
mortality discharge | 0 days after hospitalization
  To compare mortality during hospital stay in COVID-19+ patients with or without preexisting CVD.
mortality 30 days after hospitalization | 30 days after hospitalization
  To comparemortality30 days after hospital stay in COVID-19+ patients with or without preexisting CVD.
mortality 1 year after hospitalization | 1 year after hospitalization
  To compare mortality 1 year after hospital stay in COVID-19+ patients with or without preexisting CVD.

SECONDARY OUTCOMES:
Clinical outcomes according to medication at admission | 0 days after hospitalization
  Clinical outcomes according to medication at admission evaluated at hospital discharge
Clinical outcomes according to medication at admission | 30 days after hospitalization
  Clinical outcomes according to medication at admission evaluated 30 days after hospitalization
Clinical outcomes according to medication at admission | 1 year after hospitalization
  1 year after hospitalization
Clinical outcomes related to preexisting cardiovascular risk factors at admission | 0 days after hospitalization
  Clinical outcomes related to preexisting cardiovascular risk factors at admission evaluated after hospital discharge
Clinical outcomes related to preexisting cardiovascular risk factors at admission | 30 days after hospitalization
  Clinical outcomes related to preexisting cardiovascular risk factors at admission evaluated 30 days after hospital discharge
Clinical outcomes related to preexisting cardiovascular risk factors at admission | 1 year after hospitalization
  Clinical outcomes related to preexisting cardiovascular risk factors at admission evaluated 1 year after hospitalization
New onset of CVD induced by COVID-19 disease | 0 days after hospitalization
  New onset of CVD induced by COVID-19 disease at discharge
New onset of CVD induced by COVID-19 disease | 30 days after hospitalization
  New onset of CVD induced by COVID-19 disease evaluated 30 days after hospitalization
New onset of CVD induced by COVID-19 disease | 1 year after hospitalization
  New onset of CVD induced by COVID-19 disease at discharge evaluated 1 year after hospitalization
Cost of hospital stay | 0 days after hospitalization
  Cost of hospital stay
Clinical follow up at 30 days (diagnosis of new cardiac events, such as acute coronary syndromes, heart failure, arrhythmia, myocarditis). | 30 days after hospitalization
  Clinical follow up at 30 days (diagnosis of new cardiac events, such as acute coronary syndromes, heart failure, arrhythmia, myocarditis).
Clinical follow up at 1 year (diagnosis of new cardiac events, such as acute coronary syndromes, heart failure, arrhythmia, myocarditis). | 1 year after hospitalization
  Clinical follow up at 1 year (diagnosis of new cardiac events, such as acute coronary syndromes, heart failure, arrhythmia, myocarditis).

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospital (HUG), Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided